CLINICAL TRIAL: NCT02628470
Title: Effects of Cervical Manipulation and Mobilization on Salivary Cortisol Concentrations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Collaborators: Valera-Calero JA; Plaza-Manzano G; Gallego-Izquierdo T (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Dr. Pecos-Martin, D, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI/HU/2015/10
Record Dates: First submitted 2015-11-30; First posted 2015-12-11 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Neck Pain
Keywords: Cervical pain, cervicalgia
MeSH Terms: conditions — Neck Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group cervical manipulation (Experimental): The patient is supine without a pillow and physiotherapist standing in the ipsilateral corner of the hand of the thrust.
  Interventions: Procedure: cervical manipulation
- Placebo group (Placebo Comparator): Participants will receive a protocol of domiciliary cervical control exercises.
  Interventions: Procedure: cervical control exercises
- Group cervical mobilization (Active Comparator): Oscillatory mobilization technique. With the patient in prone, the investigator applies an oscillatory motion in the most painful cervical segment for three minutes
  Interventions: Procedure: Oscillatory mobilization technique

INTERVENTIONS:
Procedure: cervical manipulation — cervical high-velocity low-amplitude thrust manipulation
  Arms: group cervical manipulation
Procedure: cervical control exercises — Exercises of flexion, extension and rotation of the cervical spine
  Arms: Placebo group
Procedure: Oscillatory mobilization technique — Joint mobilization technique type III according Maitland
  Arms: Group cervical mobilization

SUMMARY:
Currently, there are many studies about the effects of manual therapy on pain, but there are not enough studies to know what are the mechanisms that cause these effects.

Although there is a research measuring neuromodulators substances after a cervical and dorsal manipulation, it has been done in healthy subjects and there is no information about mobilization. This work aims to select a sample with chronic neck pain, incorporating the cervical mobilization as a therapeutic approach to compare the effects of both techniques because not all patients accept the manipulation as a treatment technique (mobilization is much better tolerated) and to verify that the liberation of cortisol is not just caused by the stress on the joint manipulation and the psychological stress and expectation may be important.

The hypothesis of this paper is that cervical manipulation and mobilization in subjects with chronic neck pain there will increase salivary cortisol levels.

It is also expected a little increase in the expectation of being manipulated group because of the psychological stress.

It is expected an improvement in the neck disability, pain and range of motion in the intervention groups immediately after and in the three groups the following week after the exercise.

The main objective of the study is to measure and analyze changes in salivary cortisol concentrations after the intervention in the three groups. Secondary objectives is to analyze the changes in range of motion and disability caused by neck pain neck pain level

DETAILED DESCRIPTION:
STUDY DESIGN:

Experimental study using a randomized controlled trial with blinded evaluator with three parallel groups, two experimental and one placebo.

INTERVENTION

1. Experimental group cervical manipulation:

   The patient is supine without a pillow and physiotherapist standing in the ipsilateral corner of the hand of the thrust. If the segment to manipulate is the upper cervical spine, the radial aspect of the distal phalanx of the index finger of the pulse is placed on the posterolateral aspect of the transverse process of the atlas (In medium or low segments of cervical spine on the vertebra on which we want to make the thrust). The thumb rests on the zygomatic arch and the other fingers rest on the back of the skull, leaving the forearm perpendicular to the neck. In middle or lower cervical spine, the thumb rests on the angle of the jaw and the other fingers on the back of the neck.

   The contralateral hand rests against the contralateral side of the patient's skull with the fingers facing caudally, so we left ear between the index and middle fingers.

   To take the patient to the end of range of motion will be added ipsilateral inclination and contralateral rotation without exceeding the 30-40 °.

   There will be a contralateral displacement of the head and a posteroanterior glide to take the patient to energizing. The impulse is made in pure contralateral rotation.
2. Experimental Group of cervical posterior-anterior mobilization in the most painful segment:

   Maitland described by the patient is prone with his forehead in the palms. The thumb rests on the articular pillar (on the transverse blade) and the other fingers around the neck to stabilize the soft tissue.

   The limit pressure will be that cause pain to the patient. The oscillatory motion is produced by the arms and the body while the hands remain stable with a pressure distributed uniformly around the patient's neck. It is important that the neck and hands move as a unit. high-amplitude technique may be performed by raising the patient's neck with the pads of the fingers This technique was performed for 3 minutes remaining below the pain threshold of the patient.
3. Placebo group:

The subjects of this group will expect a cervical manipulation to check the psychological component has an effect on cortisol segregation. It will proceed with the same protocol as in the group of cervical manipulation, but without joint stress or thrust.

Participants will receive a protocol of domiciliary cervical control exercises adapted to each subject for deep cervical muscles after taking the second salivary sample.

Seasonal timing will be considered (evaluating the subjects in the same month), circadian rhythms (evaluating subjects mid-morning to avoid peak morning cortisol) and periods of the menstrual cycle as they are factors that can determine the results. In the case of the menstrual cycle they are cited the seventh day of the cycle.

ELIGIBILITY:
Inclusion Criteria:

* Manifest mechanical pain in the neck to the T1 vertebra as lower limit
* Present the medical diagnosis of mechanical neck pain
* Do not be getting any kind of hormonal therapy (including oral contraceptives)
* Be over 18 years old

Exclusion Criteria:

* Subjects that are associated with the adrenal gland pathology
* Pathologies excess or defect of cortisol
* Pathology severe psychological disorders related to anxiety, mood or stress
* Participants pregnant due to changes in hormonal determinations
* Contraindication to manipulation or mobilization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
salivary cortisol | Change from baseline cortisol concentration at after the intervention(immediately after)
  For measuring salivary cortisol a Cortisol kit RE52611 ELISA® will be provided by the IBL laboratory. The saliva samples will be stored at -20 ° C until analysis, being coded by the researcher and measured by a blinded assessor.
  For this, it will be added 50 uL sample of saliva in the tubes of the kit with a pipette. Subsequently 100 uL of enzyme conjugate will be added to each tube, covering the plate with adhesive and shaking carefully. It will be incubated 2 hours at room temperature (18-25 ° C) in a centrifuge at 400-600 rpm.
  After removing the adhesive and remove excess of solution wil be added 100 uL of TMB solution. It wil be centrifuged for 30 min under the same conditions. At the end, they wil be added 100 uL of TMB solution inhibitory. The results wil be measured with a photometer at 450 nm within 15 minutes of adding the last reagent.

SECONDARY OUTCOMES:
Neck Disability | Change from baseline disability at one week after intervention
  This test is a questionnaire of 10 questions to fill in the patient and disability measured by neck pain. It has been shown to have high reliability "test-retest" and be valid when compared with other measures of pain and disability
Neck pain | Change from baseline neck pain at one week after intervention
  Using a visual analogue scale (VAS) of 10 cm consisting of an opaque unnumbered rule by the front and numbered from 0 to 10 in the back side with an expression of no pain at 0 cm and maximum pain at 10 cm
Tenderness | Change from baseline pain threshold pressure at after the intervention (immediately after) and one week after
  With a algometer we will assessed the tenderness upon facet joints C2-C3 and C5-C6
Cervical joint Range | Change from baseline mobility at immediately after at one week after intervention
  Flexion, inclination, extension and rotational movement ranges will be measured with a cervical goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Tomás Gallego-Izquierdo, Dr, Study Director — Alcalá University
Locations (1):
- Alcalá Universuty, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided